CLINICAL TRIAL: NCT02654236
Title: Effect of Heavy Alcohol Consumption on Farnesoid X Receptor (FXR) Signaling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suthat Liangpunsakul (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); Intercept Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Suthat Liangpunsakul, Suthat Liangpunsakul, Associate Professor of Medicine, Biochemistry and Molecular Biology, Indiana University School of Medicine
Organization: Indiana University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: TREAT 005
Record Dates: First submitted 2016-01-06; First posted 2016-01-13 (Estimated); Results first posted 2023-04-25 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Alcohol Consumption
MeSH Terms: conditions — Alcohol Drinking | interventions — obeticholic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Heavy Drinkers on placebo
  Interventions: Drug: Placebo
- 10 mg Obeticholic Acid (OCA) (Experimental): 10 mg Obeticholic Acid (OCA) Study medication will be administered orally, once daily for 4 weeks.
  Interventions: Drug: 10 mg Obeticholic Acid (OCA)
- Non-drinking Controls (No Intervention): Non-drinking healthy controls

INTERVENTIONS:
Drug: Placebo — 1 tablet of placebo, taken orally daily with water, approximately 30 minutes prior to breakfast for 4 weeks.
  Arms: Placebo
Drug: 10 mg Obeticholic Acid (OCA) — 10 mg Obeticholic Acid (OCA) Study medication will be administered orally, once daily, approximately 30 minutes prior to breakfast for 4 weeks.
  Arms: 10 mg Obeticholic Acid (OCA)

SUMMARY:
The main purpose of this study is to see whether heavy drinking will interfere with a specific pathway, called FXR signaling in the liver. The abnormality of this pathway may lead to liver injury in some patients who drink heavily.

ELIGIBILITY:
Inclusion Criteria:

* Individuals ≥ 21 to 65 years old
* Able to provide informed consent & negative urine pregnancy test where appropriate
* Healthy controls must have not consumed any alcohol within 3 months prior to the screening visit
* Heavy alcohol drinking is defined as > 40 grams per day on average in women and > 60 grams per day on average in men for a minimum of 6 months
* Women of child bearing potential should be willing to practice contraception throughout the treatment period

Exclusion Criteria:

* Active infection as evidenced by positive urine culture, blood culture, or pneumonia
* Serum creatinine > 1.5 mg/dL
* Known co-existing infection with hepatitis C, hepatitis B, or HIV
* Significant systemic or major illness including COPD, CHF and renal failure that in the opinion of the Investigator would preclude the patient from participating in and completing the study.
* Participation in another investigational drug, biologic, or medical device trial within 30 days prior to Screening
* Previous history of jaundice or signs of liver diseases such as spider angiomata, ascites, or history of esophageal varices or hepatic encephalopathy
* Total bilirubin > 2 mg/dl and INR > 1.5 Page 20 of 37
* Women who are pregnant or nursing
* Presence of any other disease or condition that is interfering with the absorption, distribution, metabolism, or excretion of drugs including bile salt metabolism in the intestine. Patients who have undergone gastric bypass procedures will be excluded (gastric lap band is acceptable).
* Subjects who are taking warfarin

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suthat Liangpunsakul, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | 10 mg Obeticholic Acid (OCA) | Non-drinking Controls
Started | 9 | 6 | 15
Completed | 9 | 6 | 13
Not Completed | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 10 mg Obeticholic Acid (OCA) | Non-drinking Controls | Total
Number analyzed (Participants) | 9 | 6 | 15 | 30
Age, Continuous [Mean (Full Range); unit: Years] | 31 [21 to 63] | 49 [30 to 65] | 47 [27 to 60] | 39 [21 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 10 | 17
  Male | 4 | 4 | 5 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 9 | 6 | 14 | 29
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 3 | 4 | 13
  White | 3 | 2 | 7 | 12
  More than one race | 0 | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 6 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Change in Bile Salt Metabolism (C4 )Levels to Determine Effect of FXR
Time Frame: Baseline to 28 days
Population: Zero participants were analyzed due to data not being collected
Arm/Group | Placebo | 10 mg Obeticholic Acid (OCA) | Non-drinking Controls
Number analyzed (Participants) | 0 | 0 | 0

2. Primary Outcome: Change in FGF19 Levels to Determine Effect of FXR
Time Frame: Baseline to 28 days
Population: Zero participants were analyzed due to data not being collected
Arm/Group | Placebo | 10 mg Obeticholic Acid (OCA) | Non-drinking Controls
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Change in Fasting Serum Bile Salt Levels
Time Frame: Baseline to 28 days
Population: Zero participants were analyzed due to data not being collected
Arm/Group | Placebo | 10 mg Obeticholic Acid (OCA) | Non-drinking Controls
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Change in Oxidative Stress Level by Measuring Malondialdehyde
Time Frame: Baseline to 28 days
Population: Due to errors, some results were unable to be processed causing differences in the baseline and day 28.
Measure: Mean (Standard Deviation); unit: µg/ml
Arm/Group | Placebo | 10 mg Obeticholic Acid (OCA) | Non-drinking Controls
Number analyzed (Participants) | 9 | 6 | 15
µg/ml
  Baseline | 2.56 (0.79) | 2.79 (3.44) | 1.03 (1.46)
  Day 28: number analyzed (Participants) | 9 | 6 | 13
  Day 28 | 1.54 (1.77) | 3.30 (4.03) | 1.38 (0.58)

5. Secondary Outcome: Change in CYP2E1 Activity by Measuring Chlorzoxazone Clearance
Time Frame: Baseline to 28 days
Population: Zero participants were analyzed due to data not being collected
Arm/Group | Placebo | 10 mg Obeticholic Acid (OCA) | Non-drinking Controls
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Change in Gut Permeability Through Lactulose/Mannitol Test
Description: This is the measurement to quantify two non-metabolized sugar molecules-lactulose and mannitol-to determine the gut permeability
Time Frame: Baseline to 28 days
Population: Due to errors, some results were unable to be processed causing differences in the baseline and day 28.
Measure: Mean (Standard Deviation); unit: lactulose/mannitol ratio
Arm/Group | Placebo | 10 mg Obeticholic Acid (OCA) | Non-drinking Controls
Number analyzed (Participants) | 8 | 6 | 12
lactulose/mannitol ratio
  Baseline: number analyzed (Participants) | 8 | 5 | 12
  Baseline | 0.05 (0.03) | 0.04 (0.01) | 0.04 (0.02)
  Day 28: number analyzed (Participants) | 6 | 6 | 11
  Day 28 | 0.05 (0.03) | 0.07 (0.05) | 0.05 (0.05)

7. Secondary Outcome: Change in Bacterial Translocation Through Measures of Plasma LPS
Time Frame: Baseline to 28 days
Population: Due to errors, some results were unable to be processed causing differences in the baseline and day 28.
Measure: Mean (Standard Deviation); unit: Pg/ml
Arm/Group | Placebo | 10 mg Obeticholic Acid (OCA) | Non-drinking Controls
Number analyzed (Participants) | 9 | 6 | 15
Pg/ml
  Baseline | 40.22 (9.52) | 58.73 (13.3) | 58.28 (28.8)
  Day 28: number analyzed (Participants) | 9 | 6 | 13
  Day 28 | 47.84 (23.1) | 47.0 (22.3) | 19.99 (16.93)

8. Secondary Outcome: Change in Intestinal Inflammation by Measuring Stool Calprotectin
Time Frame: Baseline to 28 days
Population: Zero participants were analyzed due to data not being collected
Arm/Group | Placebo | 10 mg Obeticholic Acid (OCA) | Non-drinking Controls
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Change in Activation of Innate Immunity Through Measures of TNF-alpha
Time Frame: Baseline to 28 days
Population: Due to errors, some results were unable to be processed causing differences in the baseline and day 28.
Measure: Mean (Standard Deviation); unit: Pg/ml
Arm/Group | Placebo | 10 mg Obeticholic Acid (OCA) | Non-drinking Controls
Number analyzed (Participants) | 9 | 6 | 15
Pg/ml
  Baseline | 6.53 (3.52) | 8.99 (4.39) | 6.91 (3.36)
  Day 28: number analyzed (Participants) | 9 | 6 | 13
  Day 28 | 6.36 (3.00) | 7.97 (4.08) | 2.89 (3.27)

10. Secondary Outcome: Change in Bacterial Translocation Through Measures of Serum sCD14
Time Frame: Baseline to 28 days
Population: Due to errors, some results were unable to be processed causing differences in the baseline and day 28.
Measure: Mean (Standard Deviation); unit: µg/ml
Arm/Group | Placebo | 10 mg Obeticholic Acid (OCA) | Non-drinking Controls
Number analyzed (Participants) | 9 | 6 | 15
µg/ml
  Baseline | 2.56 (0.79) | 3.05 (0.91) | 2.09 (0.44)
  Day 28: number analyzed (Participants) | 9 | 6 | 13
  Day 28 | 2.28 (0.68) | 2.28 (0.57) | 1.38 (0.58)

11. Secondary Outcome: Change in Activation of Innate Immunity Through Measures of IL-6
Time Frame: Baseline to 28 days
Population: Zero participants were analyzed due to data not being collected
Arm/Group | Placebo | 10 mg Obeticholic Acid (OCA) | Non-drinking Controls
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Change in Activation of Innate Immunity Through Measures of IL-8
Time Frame: Baseline to 28 days
Population: Zero participants were analyzed due to data not being collected
Arm/Group | Placebo | 10 mg Obeticholic Acid (OCA) | Non-drinking Controls
Number analyzed (Participants) | 0 | 0 | 0

13. Secondary Outcome: Change in Activation of Innate Immunity Through Measures of IL-1
Time Frame: Baseline to 28 days
Population: Due to errors, some results were unable to be processed causing differences in the baseline and day 28.
Measure: Mean (Standard Deviation); unit: Pg/ml
Arm/Group | Placebo | 10 mg Obeticholic Acid (OCA) | Non-drinking Controls
Number analyzed (Participants) | 9 | 6 | 15
Pg/ml
  Baseline | 1.90 (0.28) | 1.78 (0.24) | 1.77 (0.56)
  Day 28 | 1.76 (0.32) | 1.45 (0.78) | 1.07 (0.30)

ADVERSE EVENTS:
Time Frame: Approximately 2.5 Months
Arm/Group | Placebo | 10 mg Obeticholic Acid (OCA) | Non-drinking Controls
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/6 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/6 | 0/15
Other Adverse Events (participants affected / at risk) | 4/9 | 3/6 | 0/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=9) | 10 mg Obeticholic Acid (OCA) (N=6) | Non-drinking Controls (N=15)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Burns first degree (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Thirst decreased (General disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-22): https://cdn.clinicaltrials.gov/large-docs/36/NCT02654236/Prot_SAP_000.pdf